CLINICAL TRIAL: NCT01350219
Title: Phase 2 Study of Stem Cell Educator Therapy in Type 1 Diabetes
Brief Title: Stem Cell Educator Therapy in Type 1 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Throne Biotechnologies Inc. (Industry)
Collaborators: Chinese government fundings (Unknown)
Responsible Party: Principal Investigator, Yong Zhao, MD, PhD, CEO, Throne Biotechnologies Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-037
Record Dates: First submitted 2011-05-03; First posted 2011-05-09 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes
Keywords: Cord blood stem cells; Immune modulation; Stem cell educator; Autoimmunity; Islet beta cell regeneration; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cord blood stem cell (Experimental): Human cord blood-derived multipotent stem cells (CB-SC) display unique phenotypes, such as the expression of embryonic stem (ES) cell markers, multipotential of differentiations, very low immunogenecity, and immune modulations.
  Interventions: Device: Stem Cell Educator

INTERVENTIONS:
Device: Stem Cell Educator — For the treatment, commonly the left (or right) median cubital vein, a patient's blood is passed through a Blood Cell Separator that isolates the lymphocytes from the blood according to the recommended protocol by manufacture; consequently, the collected lymphocytes were transferred into the Stem Cell Educator and treated by CB-SC; after that, the educated cells return the blood back to the patient via a dorsal vein of hand. During the MCS+ collection, the whole blood flow rate was maintained at 35 mL/min. The whole procedure was scheduled for 8 ~ 9 hrs.

SUMMARY:
The translational potential to the clinical applications of cord blood stem cells has increased enormously in recent years, mainly because of its unique advantages including no risk to the donor, no ethical issues, low risk of graft-versus-host disease (GVHD), rapid availability, and large resource worldwide. Human cord blood contains several types of stem cells such as the umbilical cord blood-derived multipotent stem cells (CB-SC). CB-SC possess multiple biological properties including the expression of embryonic stem (ES) cell characteristics, giving rise to different types of cells and immune modulation. Specifically, CB-SC can function as an immune modulator that can lead to control of the immune responses, which could in turn be used as a new approach to overcome the autoimmunity of Type 1 diabetes (T1D) in patients1 and nonobese diabetic (NOD) mice. Here, the investigators develop a novel Stem Cell Educator therapy by using CB-SC and explore the therapeutic effectiveness of Educator therapy in T1D patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients were screened for enrollment in the study if both clinical signs and laboratory tests meet the diagnosis standards of American Diabetes Association 2010. Other key inclusion criteria were presence of at least one autoantibody to the pancreatic islet β cells.

Exclusion Criteria:

* Exclusion criteria were any clinically significant diseases in liver, kidney, and heart. Additional exclusion criteria were no pregnancy, no immunosuppressive medication, no viral diseases or diseases associated with immunodeficiency.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Autoimmune control | 30 days post treatment
  Before treatment, test autoimmune-related markers as baseline; After treatment for 30 days, repeat testing autoimmune-related markers.

SECONDARY OUTCOMES:
Metabolic control | 3 months
  Before treatment, test for C-peptide levels as baseline; After treatment, test C-peptide levels on the 3rd month;
Analysis of islet beta cell function | 6 months
  1. Test for C-peptide levels on the 6th month;
  2. Full evaluation of islet beta cell function after one year.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zhao, MD, PhD, Study Chair — Throne Biotechnologies Inc.
Locations (4):
- China (3):
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - General Hospital of Jinan Military Command, Jinan, Shandong
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

REFERENCES:
- [Background] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Yin Z, Li H, Zhang Y, Diao Y, Li Y, Chen Y, Sun X, Fisk MB, Skidgel R, Holterman M, Prabhakar B, Mazzone T. Reversal of type 1 diabetes via islet beta cell regeneration following immune modulation by cord blood-derived multipotent stem cells. BMC Med. 2012 Jan 10;10:3. doi: 10.1186/1741-7015-10-3. PMID 22233865
- [Background] Zhao Y, Mazzone T. Human cord blood stem cells and the journey to a cure for type 1 diabetes. Autoimmun Rev. 2010 Dec;10(2):103-7. doi: 10.1016/j.autrev.2010.08.011. Epub 2010 Aug 20. PMID 20728583
- [Background] Zhao Y, Lin B, Darflinger R, Zhang Y, Holterman MJ, Skidgel RA. Human cord blood stem cell-modulated regulatory T lymphocytes reverse the autoimmune-caused type 1 diabetes in nonobese diabetic (NOD) mice. PLoS One. 2009;4(1):e4226. doi: 10.1371/journal.pone.0004226. Epub 2009 Jan 19. PMID 19156219
- [Background] Zhao Y. Stem cell educator therapy and induction of immune balance. Curr Diab Rep. 2012 Oct;12(5):517-23. doi: 10.1007/s11892-012-0308-1. PMID 22833322
- [Derived] Delgado E, Perez-Basterrechea M, Suarez-Alvarez B, Zhou H, Revuelta EM, Garcia-Gala JM, Perez S, Alvarez-Viejo M, Menendez E, Lopez-Larrea C, Tang R, Zhu Z, Hu W, Moss T, Guindi E, Otero J, Zhao Y. Modulation of Autoimmune T-Cell Memory by Stem Cell Educator Therapy: Phase 1/2 Clinical Trial. EBioMedicine. 2015 Nov 5;2(12):2024-36. doi: 10.1016/j.ebiom.2015.11.003. eCollection 2015 Dec. PMID 26844283
- See also: Click here for more information regarding the Stem Cell Educator therapy in clinical trials — http://www.tianhecell.com
- Available data/document: Clinical Study Report: PMC5689778 — https://www.ncbi.nlm.nih.gov/pubmed/?term=stem+cell+educator+type+1+diabetes%2C+platelets — Yong Zhao*, Zhaoshun Jiang, Elias Delgado, Heng Li, Huimin Zhou, Wei Hu, Marcos Perez-Basterrechea, Anna Janostakova, Qidong Tan, Jing Wang, Mao Mao, Zhaohui Yin, Ye Zhang, Ying Li, Quanhai Li, Jing Zhou, Yunxiang Li, Eva Martinez Revuelta, Jose Maria García-Gala, Honglan Wang, Silvia Perez-López, Maria Alvarez-Viejo, Edelmiro Menendez, Thomas Moss, Edward Guindi, Jesus Otero. Platelets-derived mitochondria display embryonic stem cell markers and improve pancreatic islet β-cell function in humans. STEM CELLS Translational Medicine. July 7, 2017. DOI: 10.1002/sctm.17-0078.